CLINICAL TRIAL: NCT04071197
Title: Gastrostomy-Biliary Diversion: Innovative Management for Children With Bile Canalicular Transport Disorders
Brief Title: Gastrostomy-Biliary Diversion: Innovative Management for Bile Canalicular Transport Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBD-PED-BCTD
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
Keywords: bile canalicular transport disorders
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Intervention Model Description: The study group will be subjected to gastrostomy followed by ERCP with nasobiliary stent placement in the CBD with its distal end been exit from the previously performed gastrostomy instead of the nostril
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrostomy-biliary tube (Experimental): The study group will be subjected to gastrostomy followed by ERCP with nasobiliary stent placement in the CBD with its distal end been exit from the previously performed gastrostomy instead of the nostril
  Interventions: Device: Gastostomy-biliary tube
- Other biliary diversion modalities (Experimental): The control group will include those cases with other modalities of therapy as external biliary diversion, internal biliary diversion, and nasobiliary tube
  Interventions: Device: External biliary diversion, internal biliary diversion and nasobiliary tube

INTERVENTIONS:
Device: Gastostomy-biliary tube — gastrostomy followed by ERCP with nasobiliary stent placement in the CBD with its distal end been exit from the previously performed gastrostomy instead of the nostril
  Arms: Gastrostomy-biliary tube
Device: External biliary diversion, internal biliary diversion and nasobiliary tube — All biliary diversion modalities other than gastrobiliary tube
  Arms: Other biliary diversion modalities

SUMMARY:
Progressive familial intrahepatic cholestasis (PFIC) is a group of disorders that can present early in life with cholestasis and intractable pruritus. Their treatment poses a great challenge, with medical treatment is not successful in many cases. Moreover, the available non-transplant surgeries carry many side effects and different degrees of efficacy. Partial external biliary diversion, internal biliary diversion, and ileal exclusion still lack widespread experience with many side effects. Nasobiliary stent placement has little tolerability, especially in younger age. Gastrobiliary tube is a novel modality for external biliary diversion in such patients.

DETAILED DESCRIPTION:
Progressive familial intrahepatic cholestasis (PFIC) is a group of disorders that can present early in life with cholestasis and intractable pruritus. They result primarily from defective transporters of different bile constituents on the canalicular membrane. The mildest form of these defective transporters can present by what is called benign recurrent intrahepatic cholestasis (BRIC).

More recently both disease categories that represent the severest (PFIC) and mildest (BRIC) forms of these transporters are better nomenclated as bile canalicular transport disorders, as some cases can start early as BRIC and later in life progress the PFIC phenotype. Moreover, a continuous spectrum of severity is present between what were previously known as PFIC and BRIC.

If the severest forms are not treated effectively they can have devastating outcomes reaching death. On the other hand, those known as BRIC can have severe attacks with unremitting pruritus that could be prolonged and sometimes persistent.

Their treatment poses a great challenge, with medical treatment is not successful in many cases. Moreover, the available non-transplant surgeries carry many side effects and different degrees of efficacy. Partial external biliary diversion is not always successful and has disfiguring effects and the stoma can have many side effects. Internal biliary diversion and ileal exclusion still lack widespread experience and encouraging results due to sometimes lack of efficacy and others due to side effects. Nasobiliary stent placement was tried in previous cases with a promising outcome, but with little tolerability, especially in younger age.

In spite liver transplant is the last resort for failing cases, the availability of successful non transplant therapy would be the preferable one if it is with adequate efficacy and little side effects. The innovative intervention proposed in this study is expected to have a good efficacy due to total biliary diversion rather than the partial ones obtained by other surgeries. Moreover, it avoids the disfiguring impact of the jeujenal stoma. More importantly, it can be removed at any time and be used at the times of severe flare of the disease.

ELIGIBILITY:
Inclusion Criteria:

* PFIC cases that are previously responding to medical treatment with recent flare of the disease that doesn't respond to medical therapy
* PFIC cases that are not responding to medical treatment and refusing non-transplant surgery and not indicated for liver transplant
* BRIC cases with frequent attacks not responding to medical therapy and refusing or unable to tolerate nasobiliary stent

Exclusion Criteria:

* Severe portal hypertensive gastropathy
* Decompensated cirrhosis

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of bleeding | 6 months
  number of patients with bleeding
Occurrence of infection | 6 months
  number of patients with infection

SECONDARY OUTCOMES:
Serum bilirubin level | 12 months
  number of patients with normal bilirubin
Improvement of pruritus | 12 months
  number of patients with no pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Sira, M.D., Principal Investigator — Pediatric Hepatology Dep; National Liver Institute, Menoufia University, Egypt
Locations (1):
- Pediatric Hepatology, Gastroenterology and Nutrition Department, National Liver Institute, Menoufia University, Shibīn al Kawm, Menofiya, Egypt

REFERENCES:
- [Background] van der Woerd WL, van Mil SW, Stapelbroek JM, Klomp LW, van de Graaf SF, Houwen RH. Familial cholestasis: progressive familial intrahepatic cholestasis, benign recurrent intrahepatic cholestasis and intrahepatic cholestasis of pregnancy. Best Pract Res Clin Gastroenterol. 2010 Oct;24(5):541-53. doi: 10.1016/j.bpg.2010.07.010. PMID 20955958
- [Background] Kaur S, Sharma D, Wadhwa N, Gupta S, Chowdhary SK, Sibal A. Therapeutic interventions in progressive familial intrahepatic cholestasis: experience from a tertiary care centre in north India. Indian J Pediatr. 2012 Feb;79(2):270-3. doi: 10.1007/s12098-011-0516-8. Epub 2011 Jul 19. PMID 21769524
- [Background] Mochizuki K, Obatake M, Takatsuki M, Nakatomi A, Hayashi T, Okudaira S, Eguchi S. Partial internal biliary diversion for patients with progressive familial intrahepatic cholestasis type 1. Pediatr Surg Int. 2012 Jan;28(1):51-4. doi: 10.1007/s00383-011-3018-x. PMID 22033772
- [Background] Stapelbroek JM, van Erpecum KJ, Klomp LW, Venneman NG, Schwartz TP, van Berge Henegouwen GP, Devlin J, van Nieuwkerk CM, Knisely AS, Houwen RH. Nasobiliary drainage induces long-lasting remission in benign recurrent intrahepatic cholestasis. Hepatology. 2006 Jan;43(1):51-3. doi: 10.1002/hep.20998. PMID 16374853